CLINICAL TRIAL: NCT06360874
Title: Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Food Effect of ND-003 Tablets in Healthy Adult Volunteers
Brief Title: A Study to Evaluate Safety, Tolerability and Pharmacokinetic of ND-003 Tablets in Healthy Adults
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen NewDEL Biotech, Co., Ltd (Industry)
Collaborators: Shenzhen Innovation Center for Small Molecule Drug Discovery Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND003-I-06
Record Dates: First submitted 2024-03-28; First posted 2024-04-11 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- ND-003 40mg (Experimental): SAD（Single Ascending Dose） Cohort 1: Participants were orally administered 40mg of ND-003 or matched placebo once.
  Interventions: Drug: ND-003 40mg; Drug: ND-003 placebo 40mg
- ND-003 80mg (Experimental): SAD Cohort 2: Participants were orally administered 80mg of ND-003 or matched placebo once.
  Interventions: Drug: ND-003 80mg; Drug: ND-003 placebo 80mg
- ND-003 160mg (Experimental): SAD Cohort 3: Participants were orally administered 160mg of ND-003 or matched placebo once.
  Interventions: Drug: ND-003 160mg; Drug: ND-003 placebo 160mg
- ND-003 240mg (Experimental): SAD Cohort 4: Participants were orally administered 240mg of ND-003 or matched placebo once.
  Interventions: Drug: ND-003 240mg; Drug: ND-003 placebo 240mg
- ND-003 300mg (Experimental): SAD Cohort 5: Participants were orally administered 300mg of ND-003 or matched placebo once.
  Interventions: Drug: ND-003 300mg; Drug: ND-003 placebo 300mg
- ND-003_Dose 1 (Experimental): MAD （Multiple Ascending Dose）Cohort 1:The dose of ND-003 or matched placebo will be determined based on the results of the SAD. Three dose cohorts will be set and the volunteers will receive the drug once a day for 7 consecutive days.
  Interventions: Drug: MAD_ND003_Dose 1; Drug: MAD_placebo_Dose 1
- ND-003_Dose 2 (Experimental): MAD Cohort 2: The dose of ND-003 or matched placebo will be determined based on the results of the SAD. Three dose cohorts will be set and the volunteers will receive the drug once a day for 7 consecutive days.
  Interventions: Drug: MAD_ND003_Dose 2; Drug: MAD_placebo_Dose 2
- ND-003_Dose 3 (Experimental): MAD Cohort 3:The dose of ND-003 or matched placebo will be determined based on the results of the SAD. Three dose cohorts will be set and the volunteers will receive the drug once a day for 7 consecutive days.
  Interventions: Drug: MAD_ND003_Dose 3; Drug: MAD_ placebo_Dose 3
- Food effect_Cohort 1 (Experimental): Food effect Cohort 1: The dose of ND-003 tablets will be determined based on the results of the SAD and MAD. Participants will be orally administered in fasting condition in day 1 and then in fed condition in day 8.
  Interventions: Drug: Food effect_Cohort 1
- Food effect_Cohort 2 (Experimental): Food effect Cohort 2: The dose of ND-003 tablets will be determined based on the results of the SAD and MAD. Participants will be orally administered in fed condition in day 1 and then in fasting condition in day 8.
  Interventions: Drug: Food effect_Cohort 2

INTERVENTIONS:
Drug: ND-003 40mg — Participants receive 40mg ND-003 tablets once.
  Arms: ND-003 40mg
Drug: ND-003 placebo 40mg — Participants receive placebo tablet matching to receive 40mg of ND-003.
  Arms: ND-003 40mg
Drug: ND-003 80mg — Participants receive 80mg ND-003 tablets once.
  Arms: ND-003 80mg
Drug: ND-003 placebo 80mg — Participants receive placebo tablet matching to receive 80mg of ND-003.
  Arms: ND-003 80mg
Drug: ND-003 160mg — Participants receive 160mg ND-003 tablets once.
  Arms: ND-003 160mg
Drug: ND-003 placebo 160mg — Participants receive placebo tablet matching to receive 160mg of ND-003.
  Arms: ND-003 160mg
Drug: ND-003 240mg — Participants receive 240mg ND-003 tablets once.
  Arms: ND-003 240mg
Drug: ND-003 placebo 240mg — Participants receive placebo tablet matching to receive 240mg of ND-003.
  Arms: ND-003 240mg
Drug: ND-003 300mg — Participants receive 300mg ND-003 tablets once.
  Arms: ND-003 300mg
Drug: ND-003 placebo 300mg — Participants receive placebo tablet matching to receive 300mg of ND-003.
  Arms: ND-003 300mg
Drug: MAD_ND003_Dose 1 — Participants will orally administrated the ND-003 tablets once a day , in which the dose will be determined based on the results of SAD.
  Arms: ND-003_Dose 1
Drug: MAD_placebo_Dose 1 — Participants will orally administrated the placebo tablets matching to the MAD_ND003_Dose 1
  Arms: ND-003_Dose 1
Drug: MAD_ND003_Dose 2 — Participants will orally administrated the ND-003 tablets once a day , in which the dose will be determined based on the results of SAD.
  Arms: ND-003_Dose 2
Drug: MAD_placebo_Dose 2 — Participants will orally administrated the placebo tablets matching to the MAD_ND003_Dose 2
  Arms: ND-003_Dose 2
Drug: MAD_ND003_Dose 3 — Participants will orally administrated the ND-003 tablets once a day , in which the dose will be determined based on the results of SAD.
  Arms: ND-003_Dose 3
Drug: MAD_ placebo_Dose 3 — Participants will orally administrated the placebo tablets matching to the MAD_ND003_Dose 3
  Arms: ND-003_Dose 3
Drug: Food effect_Cohort 1 — Firstly orally administrated ND-003 tablets in fast state and then in fed state after a 7-day washout period. Wherein, the dose will be determined based on the results of SAD and MAD.
  Arms: Food effect_Cohort 1
Drug: Food effect_Cohort 2 — Firstly orally administrated ND-003 tablets in fed state and then in fast state after a 7-day washout period. Wherein, the dose will be determined based on the results of SAD and MAD.
  Arms: Food effect_Cohort 2

SUMMARY:
The purpose of this study is to evaluate Safety, Tolerability and Pharmacokinetic of ND-003 tablets in Healthy Adults

DETAILED DESCRIPTION:
This is a Phase 1, randomized, double-blind, placebo-controlled study aimed at evaluating the safety, tolerability and Pharmacokinetic of of ND-003 in healthy adults volunteers, and then evaluate food effects.

The study will be conducted in three parts: Part A-Single ascending dose (SAD) , Part B-Multiple ascending dose (MAD) and Part C-Food Effect. Each subject will be enrolled in only one cohort of either Parts A or B or C of the study, to receive only one dose regimen during the study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Healthy volunteers, both male and female;
* 2) age: 18-45 years old;
* 3) Weight: Male ≥ 50kg, female ≥ 45kg, 19 ≤ BMI ≤ 26 (BMI=weight (kg)/height2 (m2);
* 4) Subject is in generally good health according to physical examination;
* 5) Subjects voluntarily participate in clinical trials and sign a written informed consent form.

Exclusion Criteria:

* 1) Participated in any other clinical trial of drugs within the three months prior to the trial;
* 2) Any disease that may affect the safety of the clinical trial or the in vivo process of the investigational drug;
* 3) Allergic constitution: If there is a history of drug, food allergies, or skin allergies;
* 4) Any drug that inhibits or induces liver metabolism has been used within 28 days prior to the use of the investigational drug;
* 5) Have used any medication (including Chinese herbal medicine) and health supplements within 14 days prior to administration;
* 6) Have special requirements for diet and cannot follow a unified diet;
* 7) Subjects with a history of intolerance to venipuncture blood collection, or fear of needles and hemophobia;
* 8) Drinking alcohol, tea, or caffeinated beverages for a long period of time or within 48 hours prior to administration;
* 9) Previous alcoholics, or frequent alcohol consumption within 6 months prior to administration; or consumption of any alcohol-containing product within 24 hours prior to administration ;
* 10) Blood donation or blood loss (greater than 450 mL) within 3 months prior to administration, or planning to donate blood during the study period or within 3 months after the end of the study ;
* 11) Acute illness occurred during pre study screening or prior to administration;
* 12) Subjects who have any diet that can alter liver enzymes activity within 24 hours prior to administration;
* 13) Have undergone surgery within the first three months of screening, or plan to undergo surgery during the study period;
* 14) Previous drug addict and drug abuse;
* 15) Smoking more than 5 cigarettes per day within the first 14 days of screening, or unable to withdraw nicotine-containing products during the study;
* 16) Subjects who smoke or use nicotine-containing products from screening to hospitalization;
* 17) Abnormal and clinically significant electrocardiogram results before screening or administration, or QTcF(QTcF - Fridericia's correction formula)>450 msec;
* 18) Positive results of nicotine test;
* 19) Alcohol breath test, with test results greater than 0.0mg/100 mL;
* 20) Positive urine drug test at screening;
* 21) Pregnant or lactating women;
* 22) Have plan for fertility or reluctance use any contraception during the study period and within 6 months after the end of the trial;
* 23) Subjects with other factors that are not suitable for participation in this study as judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) | through study completion, an average of 1 month
  Number and type of participants with treatment-related adverse events

SECONDARY OUTCOMES:
maximum concentration (Cmax) | Pre-dose 60 minutes and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  The drug maximum concentration reaches when the absorption rate is equal to the elimination rate at a single dose.
Time to maximum concentration (Tmax) | Pre-dose 60 minutes and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Time required to reach peak drug concentration after a single administration.
Elimination Half-life (t1/2) | Pre-dose 60 minutes and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Elimination Half-life (t1/2) refers to the time required to eliminate 50% of the drug from the body.
Clearance (CLz/F) | Pre-dose 60 minutes and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Clearance (CLz/F) describes how the body effectively eliminate drugs from the systemic circulation, typically defined as the volume of drug-containing plasma eliminated from the body per unit time.
AUC from time 0 to last time of quantifiable concentration (AUC0-t) | Pre-dose 60 minutes and 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, 96 hours post-dose
  Area under the plasma concentration-time curve from the initial administration to the last measurable concentration point.

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Shi, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei, China